CLINICAL TRIAL: NCT05374421
Title: Clinical Efficacy and Human Factors Validation Testing for Prescription Home Use of the Erchonia Corporation THL™ for Providing Relief of Tinnitus Symptoms
Brief Title: Efficacy of the Erchonia Corporation THL™ for Providing Relief of Tinnitus Symptoms
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Erchonia Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R-EAR-HOME
Record Dates: First submitted 2022-05-10; First posted 2022-05-16 (Actual); Results first posted 2024-03-12 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Tinnitus
MeSH Terms: conditions — Tinnitus

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Erchonia® THL™ (Active Comparator): The Erchonia® EVRL™ is made up of (2) 405-nanometer violet laser diodes mounted in a portable handheld device.
  Interventions: Device: Erchonia® THL™
- Placebo Laser (Placebo Comparator): The Placebo Laser has the same appearance as the Erchonia® THL™ but does not emit any therapeutic light.
  Interventions: Device: Placebo Laser

INTERVENTIONS:
Device: Erchonia® THL™ — The Erchonia® THL™ is made up of (2) 405-nanometer violet laser diodes mounted in a portable handheld device. The diodes are positioned approximately 4 inches from the skin and applied in a continuous back and forth sweeping motion from the top of the ear down the side of the neck. The treatments will be self-administered by the subject at his or her's place of residence, once per day for 28 days. Each procedure administration lasts 5 minutes per ear, for a total of 10 minutes.
  Arms: Erchonia® THL™
Device: Placebo Laser — The Placebo Laser has the same appearance as the Erchonia® THL™ but does not emit any therapeutic light. The diodes are positioned approximately 4 inches from the skin and applied in a continuous back and forth sweeping motion from the top of the ear down the side of the neck. The treatments will be self-administered by the subject at his or her's place of residence, once per day for 28 days. Each procedure administration lasts 5 minutes per ear, for a total of 10 minutes.
  Arms: Placebo Laser

SUMMARY:
The purpose of this clinical study is to determine the effectiveness of the Erchonia® THL™, manufactured by Erchonia Corporation (the Company), for prescription home use in providing relief of tinnitus symptoms when used by individuals in their own homes.

DETAILED DESCRIPTION:
Human Factors Validation Testing will initially be conducted to valuate a lay person's ability to understand and apply as applicable the information contained in the THL™ Use Device Proper Use Reference Guide, and device packaging and labeling materials to correctly, safely, and successfully activate and operate the THL™ to administer the treatment; and to identify any and all use difficulties, problems and errors, including those pertaining to critical tasks and close calls demonstrated by the lay person during device operation, and to subsequently mitigate each identified instance of use error through device and/or materials modification, and to subsequently evaluate the effectiveness of each modification, as applicable

Phase Two will commence following the successful completion of Phase One. Phase Two comprises the performance of a double-blind, randomized, placebo-controlled, clinical study of the efficacy of the Erchonia® THL™, manufactured by Erchonia Corporation (the Sponsor), for prescription home use application in providing relief of tinnitus symptoms when used by individuals in their own homes.

ELIGIBILITY:
Inclusion Criteria:

* Bilateral tinnitus
* Current diagnosis of subjective tinnitus
* No hearing loss or sensorineural hearing loss only
* 18 years of age or older
* Able to read and write English
* Constant tinnitus on-going over at least the past 6 months
* Willing to abstain from other tinnitus-related treatments, except existing hearing aid use, throughout the study duration.
* Tinnitus Functional Index (TFI) total score of 32 to 72 (Moderate to Big Problem)
* Degree of hearing loss is less than 60 dB (Moderate or less)

Exclusion Criteria:

* Tympanosclerosis
* Meniere's disease
* Acoustic neuromas
* Current and consistent use of ototoxic medications
* Presbycusis
* Thyroid disease
* Skull fracture
* Traumatic brain injury (TBI)
* Depression
* Syphilis
* Retrocochlear tumors
* Conductive hearing loss
* Pregnant, think they might be pregnant, or breastfeeding.
* Open wounds (sores, cuts, ulcers, etc) around ears or neck
* Cancerous growths around ears or neck
* Difficulty with hand dexterity sufficient to impact the ability to administer treatments with the laser such as from severe arthritis in the hands, Multiple Sclerosis, -Cerebral Palsy, Parkinson's Disease, Huntington's Disease, etc.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2022-05-10 (Actual); Primary Completion 2022-12-09 (Actual); Study Completion 2022-12-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Shanks, Study Director — Erchonia Corporation
Locations (1):
- Valley Audiology, Concord, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study procedure started with attainment of subject consent followed by subject randomization into a procedure group. Succeeding procedure group assignment the investigator performed the study qualification evaluation to determine if the subject was eligible. The "Protocol enrollment" number includes all subjects that signed the consent form, while the number of subjects that "Started" reflects the total number of subjects that satisfied the qualification criteria
Period: Overall Study
Arm/Group | Erchonia® THL™ | Placebo Laser
Started | 8 | 7
Completed | 5 | 3
Not Completed | 3 | 4
Not completed — Withdrawal by Subject | 3 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Erchonia® THL™ | Placebo Laser | Total
Number analyzed (Participants) | 8 | 7 | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 2 | 4
  >=65 years | 6 | 5 | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.4 (8.33) | 55.6 (12.25) | 64.8 (12.27)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 5 | 11
  Male | 2 | 2 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 8 | 7 | 15
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 8 | 7 | 15

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline to Study Endpoint in the Tinnitus Functional Index (TFI)
Description: The Tinnitus Functional Index (TFI) has been highly recommended to be used in both clinical and research settings for tinnitus measurement (Meikle et al., 2011). The self-report questionnaire, consists of 25 items with a response option on an 11-point Likert scale from 0-10. The calculation of overall TFI score is as follows: (1) Sum all valid answers. (2) Divide by the number of questions for which the sum of the valid answers was based to yield the respondent's mean item score. (3) Multiply by 10 to attain the respondent's overall TFI score (0-100 range). Total TFI score can be categorized as Level of Tinnitus Severity as follows: 0 to 17: Not a problem,18 to 31: Small problem, 32 to 53: Moderate problem, 54 to 72: Big Problem, 73 to 100: Very big problem.
  A negative (-) change indicates the negative impact of tinnitus on the individual's everyday life has improved (lessened).
Time Frame: Baseline and 4 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Erchonia® THL™ | Placebo Laser
Number analyzed (Participants) | 5 | 3
score on a scale | -8.96 (15.53) | -2.8 (5.7)

ADVERSE EVENTS:
Time Frame: 4 weeks
Arm/Group | Erchonia® THL™ | Placebo Laser
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/7
Other Adverse Events (participants affected / at risk) | 0/8 | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-04-13): https://cdn.clinicaltrials.gov/large-docs/21/NCT05374421/Prot_SAP_001.pdf